CLINICAL TRIAL: NCT07361822
Title: Prospective Randomized Controlled Study of Individualized PCA Model Based on Multi-dimensional Strategies (Cumulative Opioid Consumption Between Variable-Rate Feedback Infusion and Fixed-Rate Basal Infusion Modes)
Brief Title: Comparison of Cumulative Opioid Consumption Between Variable-Rate Feedback Infusion and Fixed-Rate Basal Infusion Modes of Intravenous PCA Following Mixed Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Shenzhen University General Hospital (Other); The Second Affiliated Hospital of Hainan Medical University (Other); Youjiang Medical College for Nationalities (Other); The Peoples' Hospital of Jiaozuo City (Other)
Responsible Party: Principal Investigator, Fang Luo, Director, Department of Pain Management, Principal Investigator, Clinical Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY2025-387-02-1
Record Dates: First submitted 2025-12-22; First posted 2026-01-23 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Surgery; Pain Management; Opioid Consumption; Patient-controlled Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixed-rate basal infusion mode group (Active Comparator)
  Interventions: Procedure: Fixed-rate basal infusion mode
- Variable-rate feedback infusion mode group (Experimental)
  Interventions: Procedure: Variable-rate feedback infusion mode

INTERVENTIONS:
Procedure: Fixed-rate basal infusion mode — All participants received a standardized PCA solution containing sufentanil (100 μg), ondansetron (16 mg), and normal saline with total volume 100 mL. In conventional fixed-rate basal infusion mode group, the PCA was set to administer a bolus of 2 mL with a lock out interval of 15 minutes and background infusion rate 2 mL/h.
  Arms: Fixed-rate basal infusion mode group
Procedure: Variable-rate feedback infusion mode — All participants received a standardized PCA solution containing sufentanil (100 μg), ondansetron (16 mg), and normal saline with total volume 100 mL. In variable-rate feedback infusion mode group, a bolus of 2 mL with a lock out interval of 15 minutes and background infusion rate 2 mL/h, which increased to 2.5 mL/h, was used whenever the demand dose was administered within lock out interval. The background infusion rate automatically decreased by 0.5 mL/h when the bolus button was not pressed for 1 hour. The background infusion rate was limited to a maximum of 12.0 mL/h and a minimum of 1 mL/h. The specific variable-rate feedback infusion mode setting was based on previous research, and the opinions of manufacturers and researchers to ensure patient safety and to provide effective analgesia.
  Arms: Variable-rate feedback infusion mode group

SUMMARY:
Perioperative pain management affects patient recovery. However, the rate of moderate to severe postoperative pain is as high as 73.8%, which hinders recovery and increases the risk of complications. Although opioids are the first-line analgesics, excessive use leads to adverse reactions. The traditional fixed-rate PCA mode is difficult to match the changes in postoperative pain. This study will compare different PCA mode optimization strategies, assuming that they can reduce opioid dosage, improve analgesic effect, and reduce adverse reactions, providing high-quality evidence-based basis for postoperative analgesia and promoting individualized and intelligent management.

DETAILED DESCRIPTION:
Perioperative pain management significantly impacts patient recovery outcomes. However, the incidence of moderate to severe postoperative pain remains high at 73.8%, which impedes recovery and increases complication risks. Although opioids serve as first-line analgesics, excessive use causes numerous adverse reactions. The traditional fixed-rate Patient-Controlled Analgesia (PCA) mode fails to adapt to dynamic postoperative pain variations. This study will compare different PCA optimization strategies, hypothesizing that these approaches can reduce opioid dosage, enhance analgesic effectiveness, and minimize adverse reactions. The research aims to provide evidence-based foundations for postoperative analgesia, promoting individualized and intelligent pain management systems that better serve patient needs throughout recovery.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 to 65 years;
* American Society of Anesthesiologists physical status Ⅰ - Ⅲ;
* Patients scheduled for elective mixed surgery were enrolled. Mixed surgeries included thoracoscopic surgery, laparoscopic surgery, hysteroscopy surgery, laparotomy, thoracotomy, open spinal surgery, craniotomy, and so on.

Exclusion Criteria:

* Allergy to PCA medications;
* Presence of chronic pain syndromes;
* Presence of psychiatric disorders, or severe cardiovascular, cerebrovascular, renal, or hepatic dysfunction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Estimated)
Dates: Start 2025-12-30 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Cumulative opioid consumption | Within the first 24 hours postoperatively

SECONDARY OUTCOMES:
Resting and movement pain score was assessed by NRS | At 1, 6, 12, 24, and 48 hours postoperatively
  NRS ranges from 0 to 10, with the highest score indicating the worst pain.
Cumulative PCA volume consumption | Within the first 24 hours postoperatively
Frequency of additional rescue analgesics | At 12, 24, and 48 hours postoperatively
Dosage of additional rescue analgesics | At 12, 24, and 48 hours postoperatively
Postoperative quality of recovery | At 24, and 48 hours postoperatively
  Postoperative quality of recovery was assessed through the Postoperative Quality Recovery Scale 1 day after surgery. It consists of six domains (physiologic, nociceptive, emotive, activities of daily living, cognitive and overall patient perspective). The score ranges from 0 to 150, with higher score indicating a better quality of postoperative recovery.
Quality of sleep | At 24, and 48 hours postoperatively
  Quality of sleep was evaluated on postoperative days 1, 2 and 3 using the Medical Outcomes Study Sleep Scale (MOS). MOS is questionnaire comprising 12 items that assess various aspects of sleep using a 6-point ordinal scale (1 indicating permanence and 6 indicating absence).
The level of sedation and agitation | At 12, and 24 hours postoperatively
  The level of sedation and agitation was assessed using the Richmond Agitation and Sedation Scale, which ranges from +4 (combative agitation) to -5 (deep sedation), with a score of 0 indicating an alert and calm state.
The degree of nausea and vomiting | At 12, 24, and 48 hours postoperatively
  The degree of nausea and vomiting, a score from 0 to 10 was given. A score of 0 was given if the patient had no nausea or vomiting, and a score 10 was given if the patient had severe nausea and vomiting.
The patient's satisfaction with PCA | At 24 hours postoperatively
  The patient's satisfaction with PCA during 2 days postoperatively was assessed according to the following scale: 1, very satisfactory; 2, satisfactory; 3, neutral; 4, unsatisfactory; 5; very unsatisfactory.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing 100070, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures and appendices) are available. Derived data supporting the findings of this study are available from the corresponding author Fang Luo on request.

REFERENCES:
- See also: Mitra S, Carlyle D, Kodumudi G, Kodumudi V, Vadivelu N. New Advances in Acute Postoperative Pain Management. Curr Pain Headache Rep. 2018;22(5):35. — https://pubmed.ncbi.nlm.nih.gov/29619627/
- See also: Momeni M, Crucitti M, De Kock M. Patient-controlled analgesia in the management of postoperative pain. Drugs. 2006;66(18):2321-37. — https://pubmed.ncbi.nlm.nih.gov/17181375/
- See also: Jung KT, So KY, Kim SU, Kim SH. The Optimizing Background Infusion Mode Decreases Intravenous Patient-Controlled Analgesic Volume and Opioid Consumption Compared to Fixed-Rate Background Infusion in Patients Undergoing Laparoscopic Cholecystectomy: A Pro — https://pubmed.ncbi.nlm.nih.gov/33419086/